CLINICAL TRIAL: NCT01656616
Title: Hydroxycobalamin and Rural Emergency Medical Services Cyanide Exposure Patients: A Cost Analysis
Status: Withdrawn | Type: Observational
Sponsor: MaineHealth (Other)
Responsible Party: Principal Investigator, Katrina G. Ferguson, Director of Research, Department of Emergency Medicine, MaineHealth
Other Study IDs: IRB 4053X
Record Dates: First submitted 2012-08-01; First posted 2012-08-03 (Estimated); Last update posted 2017-05-18 (Actual); Status verified 2017-05

CONDITIONS: Cyanide Poisoning
Keywords: Pharmacoeconomics; Cost effectiveness; Cyanide; Fire; Emergency Medical Services; Smoke Inhalation
MeSH Terms: conditions — Smoke Inhalation Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- EMS cyanide exposure patients
  Interventions: Drug: Cyanide antidote administration

INTERVENTIONS:
Drug: Cyanide antidote administration

SUMMARY:
The costs to a rural emergency medical services (EMS) system of a change from a traditional cyanide antidote kit to a kit containing hydroxocobalamin alone are currently unknown. The purpose of this study is to use current EMS data to calculate the costs to a rural EMS system associated with the adoption of a hydroxocobalamin protocol for the treatment of suspected cyanide exposure.

ELIGIBILITY:
Inclusion Criteria:

* Included in Maine EMS database
* House Fire Victim
* Poisoning

Exclusion Criteria:

* No potential cyanide exposure
* Incomplete data available

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: EMS patients possibly exposed to cyanide via poisoning or smoke exposure.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-08-01 (Actual); Primary Completion 2012-08-01 (Actual); Study Completion 2012-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tania D Strout, PhD, RN, MS, Study Director — MaineHealth
Locations (1):
- Maine Medical Center Department of Emergency Medicine, Portland, Maine, United States